CLINICAL TRIAL: NCT03825055
Title: Behaviour and Well-Being: A Bio-Psycho-Social Model of Resilience in Young Adults Newly Diagnosed With Multiple Sclerosis
Brief Title: Resilience in Young Adults Newly Diagnosed With Multiple Sclerosis
Acronym: BPS-ARMS
Status: Completed | Type: Observational
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other); Fondazione Italiana Sclerosi Multipla (Other); Federico II University (Other)
Responsible Party: Principal Investigator, Michela Rimondini, Associate Professor in Clinical Psychology, Universita di Verona
Other Study IDs: 2029CESC
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: disease-specific variables; biopsychosocial characteristics; resilience; adjustment; quality of life; well-being; young adults
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * blood sample (serum, whole blood)
  * sample of cerebrospinal fluid (CSF)
  * fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young patients with MS: young adults (i.e., 18-45 years) newly diagnosed with MS (Case-Only)

SUMMARY:
This study aims to fill the gap of knowledge on the biopsychosocial (BPS) characteristics and resilience of young adults newly diagnosed with Multiple Sclerosis, to evaluate the relationship among these variables, and to develop a BPS model of resilience.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is the most common neurological disease causing disability in young adults and is widely recognized as a major stress factor. Several studies have shown that the first years after the diagnosis are distressing in terms of adjustment to the disease and that MS negatively affects patients' psychological wellbeing, quality of life (QoL), and social functioning (Kern et al., 2013; Moss-Morris et al., 2013; Pagnini et al., 2014). Nevertheless, up to know, the link between disease-specific variables at diagnosis, resilience, and psychological adjustment of MS patients remains largely unexplored, especially in adolescents and young adults.

This study aims to fill the gap of knowledge on the biopsychosocial (BPS) characteristics and resilience of young adults newly diagnosed with MS, to evaluate the relationship among these variables, and to develop a BPS model of resilience.

Biological and clinical characteristics of young adults newly diagnosed with MS in the University Hospital of Verona will be investigated by collecting clinical information, performing neurological examinations, brain and cervical spinal cord magnet resonance imaging (MRI), and analyzing cerebrospinal fluid and blood biomarkers (i.e. measures of inflammation, axonal damage, oxidative stress and microRNAs (miRNAs) expression), body composition, gut microbiota, and movement/perceptual markers. Psychosocial characteristics (e.g., psychological distress, illness perception, mindfulness trait, and coping strategies), QoL, psychological wellbeing and resilience will be assessed by self-report questionnaires. Comparative statistics (i.e., ANOVA or unpaired samples t-test, correlation and regression analyses) will be applied to evaluate the relationship among biological, psychological and social factors.

The results of this study are expected not only to allow a comprehensive and new understanding of the determinants of resilience and adjustment in MS patients at this crucial stage of life but also to inform resilience interventions, tailored to adolescents' and young patients' specific needs, aiming to reduce the risk of maladaptive reactions to the disease and to improve the psychological well-being and their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* MS diagnosis in the 2 years prior to study inclusion, according to the revised McDonald Criteria (Thompson et al., 2018);
* MRI of the brain in the 6 months prior to or within one month after screening visit according to a standardized protocol (including pre- and post-contrast volumetric T1-weighted, 3D Fluid Attenuated Inversion Recovery (FLAIR), and 3D Double Inversion Recovery (DIR) sequences for brain imaging, and sagittal and axial pre- and post-contrast volumetric T1-weighted, T2-weighted and short tau inversion recovery (STIR) sequences for spinal cord imaging)
* Italian speakers.

Exclusion Criteria:

* Clinically relevant cognitive deficits as evaluated by the treating neurologist
* Treatment with any disease-modifying therapy (DMT) for MS at inclusion and by completion of study procedures (maximum two months from consent); steroids administration up to 30 days prior to inclusion is allowed.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Potentially eligible patients, diagnosed with MS in the 2 years prior to study inclusion, from the catchment area of the Multiple Sclerosis Regional Center of the Azienda Ospedaliera Universitaria Integrata of Verona will be identified during routine visits at the MS Centre of Borgo Roma Hospital Verona and asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Level of resilience | at study entry (i.e., within one month from informed consent)
  Connor-Davidson Resilience Scale (CD-RISC; Connor & Davidson, 2003), designed to assess resilience features in adolescents and adults.
  The CD-RISC is composed of 25 items and evaluated on a 5-point Likert scale (ranging from 0 "not true at all" to 4 "true nearly all of the time"), with higher scores reflecting higher levels of resilience.

SECONDARY OUTCOMES:
Level of quality of life | at study entry (i.e., within one month from informed consent)
  Italian version of the MSQOL-54 (Solari et al., 1999). The MSQOL-54 is a multidimensional health-related Quality of Life measure that combines both generic and MS-specific items, such as fatigue and cognitive function (Vickrey et al, 1995, 1997; Solari et al., 1999). The instrument generates 12 scores (physical function, role limitations-physical, role limitations-emotion, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall QoL, and sexual function) along with two summary scores (i.e., physical health and mental health) derived from a weighted combination of scale scores. There are also two single-item measures: satisfaction with sexual function and change in health.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Rimondini, PhD, Principal Investigator — Università di Verona; Alberto Gajofatto, MD, PhD, Principal Investigator — Università di Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata Verona, Policlinico G.B. Rossi, Verona, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for the primary and secondary outcome measures (resilience, quality of life) will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data can be made available upon reasonable request when data are published (6 months after publication).
Access Criteria: Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Kern S, Schrempf W, Schneider H, Schultheiss T, Reichmann H, Ziemssen T. Neurological disability, psychological distress, and health-related quality of life in MS patients within the first three years after diagnosis. Mult Scler. 2009 Jun;15(6):752-8. doi: 10.1177/1352458509103300. PMID 19482864
- [Background] Moss-Morris R, Dennison L, Landau S, Yardley L, Silber E, Chalder T. A randomized controlled trial of cognitive behavioral therapy (CBT) for adjusting to multiple sclerosis (the saMS trial): does CBT work and for whom does it work? J Consult Clin Psychol. 2013 Apr;81(2):251-62. doi: 10.1037/a0029132. Epub 2012 Jun 25. PMID 22730954
- [Background] Pagnini F, Bosma CM, Phillips D, Langer E. Symptom changes in multiple sclerosis following psychological interventions: a systematic review. BMC Neurol. 2014 Nov 30;14:222. doi: 10.1186/s12883-014-0222-z. PMID 25433519
- [Background] Solari A, Filippini G, Mendozzi L, Ghezzi A, Cifani S, Barbieri E, Baldini S, Salmaggi A, Mantia LL, Farinotti M, Caputo D, Mosconi P. Validation of Italian multiple sclerosis quality of life 54 questionnaire. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):158-62. doi: 10.1136/jnnp.67.2.158. PMID 10406981
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Vickrey BG, Hays RD, Genovese BJ, Myers LW, Ellison GW. Comparison of a generic to disease-targeted health-related quality-of-life measures for multiple sclerosis. J Clin Epidemiol. 1997 May;50(5):557-69. doi: 10.1016/s0895-4356(97)00001-2. PMID 9180648
- [Derived] Gajofatto A, Donisi V, Busch IM, Gobbin F, Butturini E, Calabrese M, Carcereri de Prati A, Cesari P, Del Piccolo L, Donadelli M, Fabene P, Fochi S, Gomez-Lira M, Magliozzi R, Malerba G, Mariotti R, Mariotto S, Milanese C, Romanelli MG, Sbarbati A, Schena F, Mazzi MA, Rimondini M. Biopsychosocial model of resilience in young adults with multiple sclerosis (BPS-ARMS): an observational study protocol exploring psychological reactions early after diagnosis. BMJ Open. 2019 Aug 2;9(8):e030469. doi: 10.1136/bmjopen-2019-030469. PMID 31377712